CLINICAL TRIAL: NCT02063269
Title: Differences of Functional Changes in Brain by Rivastigmine According to Butyrylcholinesterase Alleles in Alzheimer's Disease Patients(Rivastigmine, Imaging, and BuChE in AD: RIBA)
Brief Title: Brain Changes by Rivastigmine According to Butyrylcholinesterase Alleles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Novartis Korea Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Young Lee, MD, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CENA713DKR15T
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Alzheimer's Disease
Keywords: rivastigmine, butyrylcholinesterase, MRI, PET
MeSH Terms: conditions — Alzheimer Disease; Butyrylcholinesterase deficiency | interventions — Rivastigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rivastigmine (Experimental): Rivastigmine
  Interventions: Drug: Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine — 9-18mg/rivastigmine for 52 weeks
  Other Names: Exelon

SUMMARY:
Butyrylcholinesterase (BuChE) activity is increasing in Alzheimer Disease (AD) process (Lane et al., 2006). BuChE wild type has stronger butyrylcholine esterase activity than BuChE K variant allele and this strong activity can affect AD brain negatively by choline depletion. Rivastigmine has unique dual action - acetylcholine esterase inhibition and butyrylcholine esterase inhibition. Therefore, rivastigmine can lower serum butyrylcholine esterase activity and delay functional decrease of Fluorodeoxyglucose positron emission tomography (FDG PET) images in AD patients with BuChE wild type allele by strong BuChE inhibition.

It suggests that rivastigmine can affect brain function differently by BuChE genotype in AD. Therefore, we will try to find the different changes of serum butyrylcholine esterase activity by ELISA and functional and structural changes of brain between BuChE wild type and K-variant type by FDG PET and MRI pre and post images after 12 month use of rivastigmine.

1. Primary objective:

   1. the mean changes of Standardized Uptake Values (SUVmean) in PET imaging
   2. the mean changes of serum BuChE activity between BuChE wild type and K-variant type.
2. Secondary objectives:

   1. the mean changes of cortical thickness in brain MRI
   2. the cognitive changes in Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog)
   3. the cognitive changes in Mini-Mental State Exam (MMSE)
   4. the daily function changes by Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL)
   5. the behavioural changes by Caregiver-Administered Neuropsychiatric Inventory (NPI)
   6. the disease severity changes by Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) between BuChE wild type and K-variant type.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease (NINCD-ADRDA and MMSE between 10 ~26)
* Who didn't take Cholinesterase Inhibitor on liver within 3 months

Exclusion Criteria:

* diagnosed with diseases other than AD that affect brain atrophy according to Brain MRI
* Diagnosed with diseases other than AD which affect cognitive functions (i.g. Schizophrenia, Major Depression, Mental Retardation, encephalopathy, etc.)
* Didn't suspect of drug or alcohol addictions within last decade
* Unable to participate the study due to poor sight and hearing
* Who aren't suitable to participate according to the researchers' judgement

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
the mean changes of Standardized Uptake Values (SUVmean) in PET imaging | screening and 52weeks (2 times)
  Unit: mg/100g/min
the mean changes of serum BuChE activity between BuChE wild type and K-variant type | screening and 52weeks (2 times)
  unit of umil ACSCh/h/mg

SECONDARY OUTCOMES:
the mean changes of cortical thickness in brain MRI | screening and 52weeks (2 times)
  unit of mm
the cognitive changes in Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) | screening, 26, and 52 weeks (3 times)
  unit in points
the cognitive changes in Mini-Mental State Exam (MMSE) | screening, 26, and 52 weeks (3 times)
  unit in points
the daily function changes by Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | screening, 26, and 52 weeks (3 times)
  unit in points
the behavioural changes by Caregiver-Administered Neuropsychiatric Inventory (NPI) | screening, 26, and 52 weeks (3 times)
  unit in points
the disease severity changes by Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) between BuChE wild type and K-variant type | screening, 26, and 52 weeks (3 times)
  unit in points

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Ames A 3rd. CNS energy metabolism as related to function. Brain Res Brain Res Rev. 2000 Nov;34(1-2):42-68. doi: 10.1016/s0165-0173(00)00038-2. PMID 11086186
- [Background] Blesa R, Bullock R, He Y, Bergman H, Gambina G, Meyer J, Rapatz G, Nagel J, Lane R. Effect of butyrylcholinesterase genotype on the response to rivastigmine or donepezil in younger patients with Alzheimer's disease. Pharmacogenet Genomics. 2006 Nov;16(11):771-4. doi: 10.1097/01.fpc.0000220573.05714.ac. PMID 17047484
- [Background] Davies P, Maloney AJ. Selective loss of central cholinergic neurons in Alzheimer's disease. Lancet. 1976 Dec 25;2(8000):1403. doi: 10.1016/s0140-6736(76)91936-x. No abstract available. PMID 63862
- [Background] Fox MD, Raichle ME. Spontaneous fluctuations in brain activity observed with functional magnetic resonance imaging. Nat Rev Neurosci. 2007 Sep;8(9):700-11. doi: 10.1038/nrn2201. PMID 17704812
- [Background] Holmes C, Ballard C, Lehmann D, David Smith A, Beaumont H, Day IN, Nadeem Khan M, Lovestone S, McCulley M, Morris CM, Munoz DG, O'Brien K, Russ C, Del Ser T, Warden D. Rate of progression of cognitive decline in Alzheimer's disease: effect of butyrylcholinesterase K gene variation. J Neurol Neurosurg Psychiatry. 2005 May;76(5):640-3. doi: 10.1136/jnnp.2004.039321. PMID 15834019
- [Background] Kimura N, Kumamoto T, Masuda T, Hanaoka T, Okazaki T, Arakawa R. Evaluation of the regional cerebral blood flow changes during long-term donepezil therapy in patients with Alzheimer's disease using 3DSRT. J Neuroimaging. 2012 Jul;22(3):299-304. doi: 10.1111/j.1552-6569.2011.00612.x. Epub 2011 Jun 23. PMID 21699607
- [Background] Lane RM, Potkin SG, Enz A. Targeting acetylcholinesterase and butyrylcholinesterase in dementia. Int J Neuropsychopharmacol. 2006 Feb;9(1):101-24. doi: 10.1017/S1461145705005833. Epub 2005 Aug 5. PMID 16083515
- [Background] Levy JA, Parasuraman R, Greenwood PM, Dukoff R, Sunderland T. Acetylcholine affects the spatial scale of attention: evidence from Alzheimer's disease. Neuropsychology. 2000 Apr;14(2):288-98. doi: 10.1037//0894-4105.14.2.288. PMID 10791868
- [Background] Nobili F, Koulibaly M, Vitali P, Migneco O, Mariani G, Ebmeier K, Pupi A, Robert PH, Rodriguez G, Darcourt J. Brain perfusion follow-up in Alzheimer's patients during treatment with acetylcholinesterase inhibitors. J Nucl Med. 2002 Aug;43(8):983-90. PMID 12163621
- [Background] O'Brien KK, Saxby BK, Ballard CG, Grace J, Harrington F, Ford GA, O'Brien JT, Swan AG, Fairbairn AF, Wesnes K, del Ser T, Edwardson JA, Morris CM, McKeith IG. Regulation of attention and response to therapy in dementia by butyrylcholinesterase. Pharmacogenetics. 2003 Apr;13(4):231-9. doi: 10.1097/00008571-200304000-00008. PMID 12668920
- [Background] Poirier J. Evidence that the clinical effects of cholinesterase inhibitors are related to potency and targeting of action. Int J Clin Pract Suppl. 2002 Jun;(127):6-19. PMID 12139368
- [Background] Silverman JM, Ciresi G, Smith CJ, Marin DB, Schnaider-Beeri M. Variability of familial risk of Alzheimer disease across the late life span. Arch Gen Psychiatry. 2005 May;62(5):565-73. doi: 10.1001/archpsyc.62.5.565. PMID 15867110
- [Background] Ki CS, Na DL, Kim JW, Kim HJ, Kim DK, Yoon BK. No association between the genes for butyrylcholinesterase K variant and apolipoprotein E4 in late-onset Alzheimer's disease. Am J Med Genet. 1999 Apr 16;88(2):113-5. doi: 10.1002/(sici)1096-8628(19990416)88:23.0.co;2-3. PMID 10206226
- [Background] Kim KW, Jhoo JH, Lee JH, Lee KU, Lee DY, Youn JC, Youn JY, Woo JI. Neither the butyrylcholinesterase K variant nor transferrin C2 variant confers a risk for Alzheimer's disease in Koreans. J Neural Transm (Vienna). 2001;108(10):1159-66. doi: 10.1007/s007020170005. PMID 11725818
- [Background] Jagust WJ, Bandy D, Chen K, Foster NL, Landau SM, Mathis CA, Price JC, Reiman EM, Skovronsky D, Koeppe RA; Alzheimer's Disease Neuroimaging Initiative. The Alzheimer's Disease Neuroimaging Initiative positron emission tomography core. Alzheimers Dement. 2010 May;6(3):221-9. doi: 10.1016/j.jalz.2010.03.003. PMID 20451870